CLINICAL TRIAL: NCT05920512
Title: PLA General Hospital
Brief Title: Combination Regimen With Sodium Valproate for Severe Hemophilia: a Single-arm, Phase 1, Pilot Trial.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xue-chun Lu (Other)
Responsible Party: Sponsor-Investigator, Xue-chun Lu, Director of Hematology Department of the Second Medical Center of PLA General Hospital, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2023-261-02
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia
Keywords: Hemophilia; Sodium valproate; Sirolimus; Calcitriol
MeSH Terms: conditions — Hemophilia A | interventions — Sirolimus; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with severe haemophilia (Experimental): confirmed as hemophilia and FVIII/FIX activity <1%
  Interventions: Drug: Sodium valproate extended-release tablets

INTERVENTIONS:
Drug: Sodium valproate extended-release tablets — Sodium valproate extended-release tablets 0.5g/day; sirolimus tablets 1mg/day and calcitriol capsules 0.25μg/day.
  Other Names: sirolimus tablets; calcitriol capsules

SUMMARY:
The goal of this clinical trial is to determine the clinical efficacy and toxic effects of sodium valproate, sirolimus and calcitriol in the treatment of severe haemophilia in participants with severe haemophilia . The main questions it aims to answer are the possibility of adding a combination regimen to primary treatment for severe haemophilia . Patients will receive oral sodium valproate extended-release tablets 0.5g/day, sirolimus tablets 1mg/day and osteopontin capsules 0.25μg/day.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically confirmed severe haemophilia;
2. Expected survival of ≥ 24 weeks with an ECOG score of 0-2;
3. Not having participated in another clinical trial within four weeks;
4. Informed consent signed by the patient or an immediate family member.

Exclusion Criteria:

1. Those with other types of blood disorders diagnosed at the morphological or molecular level of the bone marrow;
2. Significantly abnormal cardiopulmonary function;
3. Hepatic or renal insufficiency;
4. Pregnancy or lactation, or inability to use contraception during the trial and for three months before the test and one year after administration
5. Persons who are allergic to the drugs likely to be used or where there is a contraindication to their use;
6. Those with severe uncontrollable infectious diseases or uncontrolled hypertension, malignancy, etc.;
7. Inability to cooperate with a regular follow-up due to psychological, social, family and other geographical circumstances;
8. Any other condition that, in the investigator's opinion, makes participation in this trial inappropriate.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
FVIII/FIX Activity | through study completion, an average of 1 month
  FVIII/FIX activity in peripheral blood
FVIII/ FIX inhibitor concentration | through study completion, an average of 1 month
  FVIII/ FIX inhibitor concentration in peripheral blood

SECONDARY OUTCOMES:
frequency of joint bleeding | through study completion, an average of 1 month
  Record the number of joint bleeds each month
Activated Partial Thromboplastin Time | through study completion, an average of 1 month
  activated partial thromboplastin time in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Xuechun Lu, M.D., Principal Investigator — Department of Hematology, the Second Medical Center of PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leissinger C. Another Victory for Patients with Hemophilia. N Engl J Med. 2023 Jan 26;388(4):372-373. doi: 10.1056/NEJMe2216176. No abstract available. PMID 36720139
- [Background] Den Uijl IE, Mauser Bunschoten EP, Roosendaal G, Schutgens RE, Biesma DH, Grobbee DE, Fischer K. Clinical severity of haemophilia A: does the classification of the 1950s still stand? Haemophilia. 2011 Nov;17(6):849-53. doi: 10.1111/j.1365-2516.2011.02539.x. Epub 2011 May 5. PMID 21545376
- [Background] DiMichele D. Inhibitor development in haemophilia B: an orphan disease in need of attention. Br J Haematol. 2007 Aug;138(3):305-15. doi: 10.1111/j.1365-2141.2007.06657.x. PMID 17614818
- [Background] Jankowska KI, McGill J, Pezeshkpoor B, Oldenburg J, Atreya CD, Sauna ZE. Clinical manifestation of hemophilia A in the absence of mutations in the F8 gene that encodes FVIII: role of microRNAs. Transfusion. 2020 Feb;60(2):401-413. doi: 10.1111/trf.15605. Epub 2019 Nov 29. PMID 31785023
- [Background] Marchesini E, Morfini M, Valentino L. Recent Advances in the Treatment of Hemophilia: A Review. Biologics. 2021 Jun 15;15:221-235. doi: 10.2147/BTT.S252580. eCollection 2021. PMID 34163136
- [Background] Lu P, Yan M, He L, Li J, Ji Y, Ji J. Crosstalk between Epigenetic Modulations in Valproic Acid Deactivated Hepatic Stellate Cells: An Integrated Protein and miRNA Profiling Study. Int J Biol Sci. 2019 Jan 6;15(1):93-104. doi: 10.7150/ijbs.28642. eCollection 2019. PMID 30662350
- [Background] Moghimi B, Sack BK, Nayak S, Markusic DM, Mah CS, Herzog RW. Induction of tolerance to factor VIII by transient co-administration with rapamycin. J Thromb Haemost. 2011 Aug;9(8):1524-33. doi: 10.1111/j.1538-7836.2011.04351.x. PMID 21585650
- [Background] Johannessen SI, Landmark CJ. Antiepileptic drug interactions - principles and clinical implications. Curr Neuropharmacol. 2010 Sep;8(3):254-67. doi: 10.2174/157015910792246254. PMID 21358975
- [Background] Mintzer S, Mattson RT. Should enzyme-inducing antiepileptic drugs be considered first-line agents? Epilepsia. 2009 Sep;50 Suppl 8:42-50. doi: 10.1111/j.1528-1167.2009.02235.x. PMID 19702733
- [Background] Verrotti A, Coppola G, Parisi P, Mohn A, Chiarelli F. Bone and calcium metabolism and antiepileptic drugs. Clin Neurol Neurosurg. 2010 Jan;112(1):1-10. doi: 10.1016/j.clineuro.2009.10.011. Epub 2009 Nov 12. PMID 19913352
- [Result] Stanford S, Pink R, Creagh D, Clark A, Lowe G, Curry N, Pasi J, Perry D, Fong S, Hayes G, Chandrakumaran K, Rangarajan S. Adenovirus-associated antibodies in UK cohort of hemophilia patients: A seroprevalence study of the presence of adenovirus-associated virus vector-serotypes AAV5 and AAV8 neutralizing activity and antibodies in patients with hemophilia A. Res Pract Thromb Haemost. 2019 Jan 25;3(2):261-267. doi: 10.1002/rth2.12177. eCollection 2019 Apr. PMID 31011710
- [Result] Nathwani AC, Gray JT, McIntosh J, Ng CY, Zhou J, Spence Y, Cochrane M, Gray E, Tuddenham EG, Davidoff AM. Safe and efficient transduction of the liver after peripheral vein infusion of self-complementary AAV vector results in stable therapeutic expression of human FIX in nonhuman primates. Blood. 2007 Feb 15;109(4):1414-21. doi: 10.1182/blood-2006-03-010181. Epub 2006 Nov 7. PMID 17090654
- [Result] Mingozzi F, Anguela XM, Pavani G, Chen Y, Davidson RJ, Hui DJ, Yazicioglu M, Elkouby L, Hinderer CJ, Faella A, Howard C, Tai A, Podsakoff GM, Zhou S, Basner-Tschakarjan E, Wright JF, High KA. Overcoming preexisting humoral immunity to AAV using capsid decoys. Sci Transl Med. 2013 Jul 17;5(194):194ra92. doi: 10.1126/scitranslmed.3005795. PMID 23863832
- [Result] Puetz J, Soucie JM, Kempton CL, Monahan PE; Hemophilia Treatment Center Network (HTCN) Investigators. Prevalent inhibitors in haemophilia B subjects enrolled in the Universal Data Collection database. Haemophilia. 2014 Jan;20(1):25-31. doi: 10.1111/hae.12229. Epub 2013 Jul 16. PMID 23855900
- [Result] Rocca A, Minucci S, Tosti G, Croci D, Contegno F, Ballarini M, Nole F, Munzone E, Salmaggi A, Goldhirsch A, Pelicci PG, Testori A. A phase I-II study of the histone deacetylase inhibitor valproic acid plus chemoimmunotherapy in patients with advanced melanoma. Br J Cancer. 2009 Jan 13;100(1):28-36. doi: 10.1038/sj.bjc.6604817. PMID 19127265
- [Result] Nilubol N, Merkel R, Yang L, Patel D, Reynolds JC, Sadowski SM, Neychev V, Kebebew E. A phase II trial of valproic acid in patients with advanced, radioiodine-resistant thyroid cancers of follicular cell origin. Clin Endocrinol (Oxf). 2017 Jan;86(1):128-133. doi: 10.1111/cen.13154. Epub 2016 Sep 8. PMID 27392538
- [Result] Nathwani AC, Tuddenham EG, Rangarajan S, Rosales C, McIntosh J, Linch DC, Chowdary P, Riddell A, Pie AJ, Harrington C, O'Beirne J, Smith K, Pasi J, Glader B, Rustagi P, Ng CY, Kay MA, Zhou J, Spence Y, Morton CL, Allay J, Coleman J, Sleep S, Cunningham JM, Srivastava D, Basner-Tschakarjan E, Mingozzi F, High KA, Gray JT, Reiss UM, Nienhuis AW, Davidoff AM. Adenovirus-associated virus vector-mediated gene transfer in hemophilia B. N Engl J Med. 2011 Dec 22;365(25):2357-65. doi: 10.1056/NEJMoa1108046. Epub 2011 Dec 10. PMID 22149959
- [Result] Rangarajan S, Walsh L, Lester W, Perry D, Madan B, Laffan M, Yu H, Vettermann C, Pierce GF, Wong WY, Pasi KJ. AAV5-Factor VIII Gene Transfer in Severe Hemophilia A. N Engl J Med. 2017 Dec 28;377(26):2519-2530. doi: 10.1056/NEJMoa1708483. Epub 2017 Dec 9. PMID 29224506